CLINICAL TRIAL: NCT02649582
Title: Adjuvant Dendritic-Cell Immunotherapy Plus Temozolomide Following Surgery and Chemoradiation in Patients With Newly Diagnosed Glioblastoma
Brief Title: Adjuvant Dendritic Cell-immunotherapy Plus Temozolomide in Glioblastoma Patients
Acronym: ADDIT-GLIO
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Zwi Berneman, Full Professor, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCRG14-001
Record Dates: First submitted 2015-01-23; First posted 2016-01-07 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Glioblastoma Multiforme of Brain
Keywords: Dendritic cells; Chemoimmunotherapy; Adjuvant therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Dendritic cell vaccine plus temozolomide chemotherapy
  Interventions: Biological: Dendritic cell vaccine plus temozolomide chemotherapy

INTERVENTIONS:
Biological: Dendritic cell vaccine plus temozolomide chemotherapy — When eligible after total or subtotal resection (as assessed by neurosurgeon and post-operative brain MRI):
  1. Leukocyte apheresis (before chemoradiation): for DC vaccine production
  2. Chemoradiation (standard treatment: initiated as soon as the patient's hematological blood values are adequate after apheresis): 2 Gy once daily 5 days/week for 6 weeks with 75 mg/m² temozolomide daily from the first until the last day of radiotherapy (no longer than 49 days in total)
  3. Induction immunotherapy: intradermal vaccination with autologous WT1 mRNA-loaded DCs weekly (+/-1 day) for 3 weeks, starting ≥ 1 week after radiotherapy
  4. Chemo-immunotherapy: 150-200 mg/m²/d temozolomide days 1-5 every 28 days +/- 2 days (max. 12 months) starting ≥3 days after the third vaccine of the induction immunotherapy + DC vaccination on day 21±3 days of every 28-day cycle

SUMMARY:
In this phase I/II trial, the primary objective is to determine overall and progression-free survival of patients with newly diagnosed glioblastoma when autologous Wilms' tumor 1 (WT1) messenger (m)RNA-loaded dendritic cell (DC) vaccination is added to adjuvant temozolomide maintenance treatment following (sub)total resection and temozolomide-based chemoradiation.

DETAILED DESCRIPTION:
Glioblastoma multiforme (GBM), a microscopically infiltrative disease, is the most common malignant brain tumor worldwide. Despite optimized standard of care treatment median survival and prognosis remain poor with a median survival of only 15% and five year survival after diagnosis of 5%.

In this single arm single centre phase I/II trial the investigators will determine the overall and progression free survival of patients with newly diagnosed GBM when autologous WT1 mRNA loaded dendritic cell vaccination is added to standard of care treatment. During recruitment, the investigators will include 20 patients with newly diagnosed, histologically verified glioblastoma (WHO grade IV) who have received a total or subtotal resection of the tumor. Patients who underwent prior radiation or chemotherapy or with a history of other malignancy will be excluded. In addition to standard of care consisting of adjuvant chemoradiation with temozolomide and temozolomide maintenance patients will receive an intradermal vaccination with autologous WT1 mRNA-loaded dendritic cells commencing 1 week after radiotherapy. The dendritic cell therapy product will be generated and administered in the Antwerp University Hospital, more specifically the Center for Cell Therapy and Regenerative Medicine (CCRG), headed by Prof. Zwi Berneman and the Division of Hematology.

Recruitment began in December 2015 and is intended to continue until the end of 2024 or when 20 patients are enrolled. After a follow-up period (until 90 days after final DC vaccine administration or 24 months after apheresis , whichever occurs later), overall and progression free survival analysis will be performed and this will be compared with the published data of standard of care treatment without vaccination. In addition the investigators will look for feasibility, incidence of adverse events and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histologically verified glioblastoma (WHO grade IV)
* Aged ≥ 18 years
* Total or subtotal resection:

  * Total resection: macroscopic complete resection as assessed by the neurosurgeon and absence of any residual contrast-enhancing mass on post-operative (≤ 72h) brain MRI
  * Subtotal resection: macroscopic complete resection as assessed by the neurosurgeon, but with residual contrast-enhancement ≤ 2 cm³ on post-operative (≤ 72h) brain MRI
* Signed informed consent
* Willing and able to comply with the protocol as judged by the Investigator
* Estimated to start with chemoradiation ≥ 28 days and ≤ 49 days following surgical resection
* Fit to undergo: leukapheresis, chemoradiation, chemotherapy and immunotherapy
* No corticosteroid treatment ≤ 1 week before apheresis
* WHO performance status ≤ 2
* Life expectancy ≥ 3 months as estimated by the Investigator

Exclusion Criteria:

* History of another malignancy, except for adequately controlled basal cell skin carcinoma, squamous skin carcinoma, or carcinoma in situ of the uterine cervix or unless the investigator rationalizes otherwise
* Prior radiation or chemotherapy
* Any pre-existing contraindication for temozolomide treatment
* Any pre-existing contraindication for contrast-enhanced brain MRI
* Pregnant or breast-feeding
* Documented immune deficiency or systemic immune-suppressive treatment
* Known positive viral serology for HIV, HBV, HCV, or syphilis
* Any other condition, either physical or psychological, or reasonable suspicion thereof on clinical or special investigation, which contraindicates the use of the vaccine, or may negatively affect patient compliance, or may place the patient at higher risk of potential treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Through study completion with follow-up until 90 days after final DC vaccine administration or 24 months after apheresis, whichever occurs later
  Patients will be followed for survival, from apheresis (~ diagnosis), for which the accurate date and reason of death (cancer-related or non-related) will be recorded for every patient.

SECONDARY OUTCOMES:
Number of glioblastoma patients post surgical resection with feasible and safe DC vaccine production | Vaccine production and quality testing (i.e. 4 weeks after leukapheresis)
  Production of autologous DC vaccines from newly diagnosed glioblastoma patients that underwent maximal, safe surgical resection will be evaluated for:
  1. feasibility, assessed by success of leukapheresis and production of sufficient and qualified (phenotypic and functional requirements) vaccines.
  2. Safety, assessed by microbiological testing (bacteria, yeast, fungi, mycoplasma, endotoxin) of the DC vaccines.
Feasibility of DC vaccine administration to glioblastoma patients combined with chemotherapy | Upon maintenance chemotherapy treatment (i.e. +/- 12 weeks post leukapheresis)
  Administration of 3 weekly DC vaccines following adjuvant chemoradiation (induction phase) and additional DC vaccination at day 21 of each maintenance chemotherapy cycle (booster phase) will be evaluated for feasibility, assessed by successful DC vaccine administration of the proposed treatment scheme.
Number of participants with adverse events as a measure of safety and tolerability | Through study completion with follow-up until 90 days after final DC vaccine administration or 24 months after apheresis, whichever occurs later
  Monitoring the incidence of adverse events to evaluate the safety profile and tolerability of the treatment. The severity of adverse events will be assessed according to the NCI CTCAE scale (v4.03, published June 14, 2010).
Immunological responses to the DC vaccine | At first DC vaccination + day 1 of first and fourth temozolomide treatment cycles
  Immunological responses to the vaccine will be evaluated ex vivo. Blood samples will be collected from patients on the day of the first DC vaccine, and on day 1 of the first and fourth maintenance temozolomide treatment cycles and will be examined for cell subset distribution and activation status and antigen-specific immunity.
Objective clinical responses by tumor evaluation (clinical efficacy) | Through study completion with follow up until 90 days after final DC vaccine administration or 24 months after apheresis, whichever occurs later
  Disease evolution and progression-free survival will be assessed according to the Response Assessment in Neuro-Oncology (RANO) criteria, based on imaging findings (MRI, CT), clinical status and corticosteroid use.
  Disease will be assessed following chemoradiation (≤ 2 weeks after completing chemoradiation), after every two cycles of temozolomide maintenance treatment and at least every 12 weeks during the booster phase, and every 9-12 weeks during follow-up after treatment discontinuation.

OTHER OUTCOMES:
General and disease-specific quality of life | Through study completion with follow up until 90 days after final DC vaccine administration or 24 months after apheresis, whichever occurs later
  Patients will be asked to fill out general and disease-specific quality of life questionnaires to assess changes in general and disease-specific quality of life during the study at regular time points.

CONTACTS AND LOCATIONS:
Overall Officials: Zwi N Berneman, MD, PhD, Study Director — Antwerp University Hospital, Division of Hematology and Center for Cell Therapy and Regenerative Medicine; Marika Rasschaert, MD, PhD, Principal Investigator — Antwerp University Hospital (UZA), Division of Oncology
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

REFERENCES:
- [Background] Van Tendeloo VF, Van de Velde A, Van Driessche A, Cools N, Anguille S, Ladell K, Gostick E, Vermeulen K, Pieters K, Nijs G, Stein B, Smits EL, Schroyens WA, Gadisseur AP, Vrelust I, Jorens PG, Goossens H, de Vries IJ, Price DA, Oji Y, Oka Y, Sugiyama H, Berneman ZN. Induction of complete and molecular remissions in acute myeloid leukemia by Wilms' tumor 1 antigen-targeted dendritic cell vaccination. Proc Natl Acad Sci U S A. 2010 Aug 3;107(31):13824-9. doi: 10.1073/pnas.1008051107. Epub 2010 Jul 14. PMID 20631300
- [Background] Van Driessche A, Van de Velde AL, Nijs G, Braeckman T, Stein B, De Vries JM, Berneman ZN, Van Tendeloo VF. Clinical-grade manufacturing of autologous mature mRNA-electroporated dendritic cells and safety testing in acute myeloid leukemia patients in a phase I dose-escalation clinical trial. Cytotherapy. 2009;11(5):653-68. doi: 10.1080/14653240902960411. PMID 19530029
- [Background] Van Driessche A, Berneman ZN, Van Tendeloo VF. Active specific immunotherapy targeting the Wilms' tumor protein 1 (WT1) for patients with hematological malignancies and solid tumors: lessons from early clinical trials. Oncologist. 2012;17(2):250-9. doi: 10.1634/theoncologist.2011-0240. Epub 2012 Jan 30. PMID 22291091
- [Background] Smits EL, Anguille S, Cools N, Berneman ZN, Van Tendeloo VF. Dendritic cell-based cancer gene therapy. Hum Gene Ther. 2009 Oct;20(10):1106-18. doi: 10.1089/hum.2009.145. PMID 19656053
- [Background] Anguille S, Smits EL, Lion E, van Tendeloo VF, Berneman ZN. Clinical use of dendritic cells for cancer therapy. Lancet Oncol. 2014 Jun;15(7):e257-67. doi: 10.1016/S1470-2045(13)70585-0. PMID 24872109
- [Background] Anguille S, Smits EL, Bryant C, Van Acker HH, Goossens H, Lion E, Fromm PD, Hart DN, Van Tendeloo VF, Berneman ZN. Dendritic Cells as Pharmacological Tools for Cancer Immunotherapy. Pharmacol Rev. 2015 Oct;67(4):731-53. doi: 10.1124/pr.114.009456. PMID 26240218
- [Background] Willemen Y, Huizing MT, Smits E, Anguille S, Nijs G, Stein B, Van Tendeloo V, Peeters M, Berneman Z. J Clin Oncol 30(suppl): abstr e13051, 2012.
- [Background] Anguille S, Van de Velde AL, Smits EL, Van Tendeloo VF, Juliusson G, Cools N, Nijs G, Stein B, Lion E, Van Driessche A, Vandenbosch I, Verlinden A, Gadisseur AP, Schroyens WA, Muylle L, Vermeulen K, Maes MB, Deiteren K, Malfait R, Gostick E, Lammens M, Couttenye MM, Jorens P, Goossens H, Price DA, Ladell K, Oka Y, Fujiki F, Oji Y, Sugiyama H, Berneman ZN. Dendritic cell vaccination as postremission treatment to prevent or delay relapse in acute myeloid leukemia. Blood. 2017 Oct 12;130(15):1713-1721. doi: 10.1182/blood-2017-04-780155. Epub 2017 Aug 22. PMID 28830889
- [Background] Z. Berneman, A. Van de Velde, S. Anguille, Y. Willemen, M. Huizing, P. Germonpré, K. Saevels, G. Nijs, N. Cools, A. Van Driessche, B. Stein, H. De Reu, W. Schroyens, A. Gadisseur, A. Verlinden, K. Vermeulen, M. Maes, M. Lammens, H. Goossens, M. Peeters, V. Van Tendeloo, E. Smits. Vaccination with Wilms' Tumor Antigen (WT1) mRNA-Electroporated Dendritic Cells as an Adjuvant Treatment in 60 Cancer Patients: Report of Clinical Effects and Increased Survival in Acute Myeloid Leukemia, Metastatic Breast Cancer, Glioblastoma and Mesothelioma. Cytotherapy 2016, 18(6), p. S13-14
- [Background] Z. Berneman, S. Anguille, Y. Willemen, A. Van de Velde, P. Germonpré, M. Huizing, V. Van Tendeloo, K. Saevels, L. Rutsaert, K. Vermeulen, A. Snoeckx, B. Op de Beeck, N. Cools, G. Nijs, B. Stein, E. Lion, A. van Driessche, M. Peeters, E. Smits. Vaccination of cancer patients with dendritic cells electroporated with mRNA encoding the Wilms' Tumor protein (WT1): correlation of clinical effect and overall survival with T-cell response. Cytotherapy 2019, 21(5), p. S10.